CLINICAL TRIAL: NCT06967779
Title: Analysis of the Relationship Between the Concentration of the Brain Derived Neurotrophic Factor (BDNF) in Plasma, the Occurrence of BDNF Gene Polymorphism (Val66Met) and White Blood Cell Markers and the Incidence of Postoperative Central Nervous System Disorders in Patients Undergoing General Anesthesia for Cardiac Surgery With Extracorporeal Circulation
Brief Title: The Relationship Between Delirium and BDNF in Coronary Artery Bypass Graft Surgery
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Kacper Lechowicz, PhD student, Pomeranian Medical University Szczecin
Other Study IDs: delirium CABG
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Delirium - Postoperative; BDNF; CABG
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is aimed at finding a correlation between postoperative delirium occurrence, severity and duration after cardiac surgery and the level of brain-derived neurotrophic factor (BDNF) in plasma as a marker of brain injury induced by cardio-pulmonary by-pass and its association with genetic predisposition in patients undergoing coronary artery bypass grafting (CABG) carrying BDNF gene polymorphism (Val66Met).

ELIGIBILITY:
Inclusion criteria include:

1. Age > 18 years.
2. Planned coronary artery bypass grafting (CABG) procedure with the use of cardiopulmonary by-pass (CPB).
3. Ability to understand and sign an informed consent form.

Exclusion criteria include:

1. Emergency surgery.
2. Previous known cognitive disorders: Mini Mental State Examination (MMSE) score <15.
3. Baseline delirium (positive CAM test prior to surgery).
4. Diagnosis of psychiatric syndromes in the past - i.e. depression, dementia, psychosis or schizophrenia.
5. Inability to understand Polish language.
6. Inability to give and sign informed consent due to auditory or visual dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective observational cohort study will recruit 200 patients scheduled for planned coronary artery bypass grafting (CABG), with the use of cardio-pulmonary by-pass who will be operated at the Cardiac Surgery Department of the Pomeranian Medical University in Szczecin. The Cardiac Surgery Department of Pomeranian Medical University has a volume of 900-1100 operations per year, 70% being CABG (approx. 700 CABG operations per year).
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The main aim of the study will be to assess the correlation between brain function disorders, defined as abnormal BDNF levels, and postoperative delirium. | Up to a year after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersytecki Szpital Kliniczny nr 2 PUM w Szczecinie, Szczecin, West Pomeranian Voivodeship, Poland